CLINICAL TRIAL: NCT06637293
Title: Deployment and Evaluation of Artificial Intelligence Software for Electrocardiogram Analysis and Management in Primary Care
Acronym: DAISEA-ECG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Robert Avram, Interventional cardiologist, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DAISEA-ECG
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Primary Care Provider; Structural Heart Disease

STUDY DESIGN:
Intervention Model Description: stepped wedge randomization
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No DeepECG plateform diagnosis & recommendations (No Intervention)
- DeepECG plateform diagnosis & recommendations (Experimental)
  Interventions: Device: DeepECG plateform diagnosis & recommendations

INTERVENTIONS:
Device: DeepECG plateform diagnosis & recommendations — EchoNeXT& ECG-AI algorithm
  Arms: DeepECG plateform diagnosis & recommendations

SUMMARY:
The DAISEA-ECG project aims to improve the diagnosis of heart diseases in primary care through the DeepECG platform, which combines ECG-AI and ECHONeXT algorithms. This study uses a stepped wedge design, where each Family Medicine Group acts as its own control. The FMGs will gradually transition from the control period (without AI recommendations) to the intervention period (with AI recommendations activated) in a randomized sequence.

The primary objective is to compare the sensitivity of family physicians in detecting cardiac pathologies, with and without the assistance of the DeepECG platform. Sensitivity is defined as the proportion of patients correctly referred to cardiology or for transthoracic echocardiography (TTE) among those who indeed required cardiovascular evaluation, as confirmed by an independent adjudication committee.

DETAILED DESCRIPTION:
Mathematically, sensitivity is calculated as True Positive / (True Positive + False Negative), where True Positive represents correctly referred patients and false negatives represents patients who should have been referred but were not.

The secondary objectives include determining the rate of cardiovascular evaluation referrals before and after the intervention (implementation of the DeepECG platform), the individual characteristics of the intervention (PPV, NPV, and specificity), as well as evaluating the feasibility of implementing AI-based automatic ECG interpretation in primary care through surveys of family physicians and cardiologists.

PPV: Positive predictive value NPV: Negative predictive value

ELIGIBILITY:
Inclusion Criteria:

Family Physicians or Nurse Practitioners

Family physicians or nurse practitioners (NPs) practicing in one of the participating FMGs.

Family physicians who have given their free and informed consent. Patients

Adult patients (18 years or older). Patients without follow-up in cardiology or internal medicine for cardiovascular issues (arrhythmia, heart failure, myocardial infarction, atherosclerotic coronary artery disease, valvular heart disease) or those who had a negative investigation in the past with no additional follow-up.

ECG

Any 12-lead ECG performed with the MUSE GE 360 machine. ECG of adequate technical quality for interpretation (otherwise, it will be automatically rejected by the platform).

-

Exclusion Criteria:

* Family Physicians or Nurse Practitioners

Family physicians practicing exclusively in pediatrics (patients under 18 years old).

Family physicians unable to follow the project guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
sensitivity of cardiology referrals | 18 months
  Compare the sensitivity of cardiology referrals made by family physicians and nurse practitioners before and after the activation of AI-assisted diagnostics and recommendations from the DeepECG platform.

SECONDARY OUTCOMES:
specificity, negative predictive value, and positive predictive value of cardiology referrals | 18 months
  Compare the specificity, negative predictive value, and positive predictive value of cardiology referrals made by family physicians and nurse practitioners before and after the activation of AI-assisted diagnostics and recommendations.

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.heartwise.ai/